CLINICAL TRIAL: NCT02586376
Title: Effects of the Different Intensities of the Low-level Laser Therapy on Handgrip Test on Patients With Kidneys Failure: A Randomized, Controlled Clinical Trail
Brief Title: Effects of the Low-level Laser Therapy (LLLT) on Muscle Strength (MS) of the Patients With Kidneys Failure (KF)
Acronym: LLLTMSKF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Fabrício Edler Macagnan, Clinical Research, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: LLLT-RENAIS-2015
Record Dates: First submitted 2015-10-05; First posted 2015-10-26 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Kidney Failure
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0J LLLT (Sham Comparator): The intervention will be made with the machine off.
  Interventions: Device: 0J LLLT
- 4J LLLT (Experimental): The Laser radiation will be made with 4J by spot.
  Interventions: Device: 4J LLLT
- 6J LLLT (Experimental): The Laser radiation will be made with 6J by spot.
  Interventions: Device: 6J LLLT
- 8J LLLT (Experimental): The Laser radiation will be made with 8J by spot.
  Interventions: Device: 8J LLLT

INTERVENTIONS:
Device: 0J LLLT — Sham Low-Level Laser Therapy (Sham LLLT): perform with the machine off.
  Other Names: Sham LLLT
  Arms: 0J LLLT
Device: 4J LLLT — 4J Low-Level Laser Therapy (4J LLLT) irradiation will be perform with 4J.
  Other Names: 4J
  Arms: 4J LLLT
Device: 6J LLLT — 6J Low-Level Laser Therapy (6J LLLT) irradiation will be perform with 6J.
  Other Names: 6J
  Arms: 6J LLLT
Device: 8J LLLT — 8J Low-Level Laser Therapy (8J LLLT) irradiation will be perform with 8J.
  Other Names: 8J
  Arms: 8J LLLT

SUMMARY:
The low-level laser therapy (LLLT) has been used in many inflammatory disorders. More recently the LLLT was associated with an improvement in the muscle strength and endurance. But, these effects were described only in health or athletic individuals. In this randomized and controlled clinical trails, the investigators will study the effects of LLLT on muscle strength of the patients with kidneys failure on long time hemodialysis treatment. Additionally, investigators will explore three different intensities up the muscle strength.

DETAILED DESCRIPTION:
This study will be conducing in a large hospital that is reference in kidneys disorders treatments. 16 patients will be randomized for placebo, 4J, 6J, or 8J low-level laser therapy (LLLT). The maximal voluntary contraction (MVC) will be test by handgrip test before and after de LLLT. One-week interval between the LLLT will gave to reduce the influence between the treatments. Moreover the endurance test will be use to evaluate the muscle oxidation impact of the LLLT.

ELIGIBILITY:
Inclusion Criteria:

* chronic kidney failure,
* long time hemodialysis treatment (>18 months)

Exclusion Criteria:

* any health disturbance that can reduces the handgrip test performance beyond to the produced by the chronic kidney failure.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-10; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Muscle Strength (Handgrip Test) | once a week throughout 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fabrício E. Macagnan, PhD, Principal Investigator — Universidade Federal de Ciências da Saúde
Locations (1):
- Fabrício Edler Macagnan, Porto Alegre, Rio Grande do Sul, Brazil